CLINICAL TRIAL: NCT05806814
Title: Pilot Trial to Investigate Immune Response to an Extended Course of Sipuleucel-T Immunotherapy in Patients With Metastatic Castration-resistant Prostate Cancer (OU-SCC-EXCITE)
Brief Title: Sipuleucel-T Based Autologous Cellular Immunotherapy for Advanced Prostate Cancer
Acronym: OU-SCC-EXCITE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Dendreon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OU-SCC-EXCITE
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Keywords: antigen presenting cells (APCs); Sipuleucel-T (Sip-T); granulocyte-macrophage colony-stimulating factor (GM-CSF); prostatic acid phosphatase (PAP)
MeSH Terms: interventions — sipuleucel-T

STUDY DESIGN:
Intervention Model Description: The primary objective is to evaluate the feasibility and immune response of an extended course of Sipuleucel-T immunotherapy given at week 0, 2, and 12-14 in patients with metastatic castration-resistant prostate cancer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Extended course of Sipuleucel-T treatment (Experimental)
  Interventions: Biological: Sipuleucel-T

INTERVENTIONS:
Biological: Sipuleucel-T — Three doses of Sipuleucel-T, each containing a minimum of 50 million autologous CD54+ cells activated with PAP-GM-CSF, given at week 0, 2, and 12-14.
  Other Names: PROVENGE

SUMMARY:
Proposed immunotherapy with an extended course of Sipuleucel-T treatment may induce a more robust immune response and improve the anti-cancer efficacy of Sipuleucel-T in patients with metastatic Castration-Resistant Prostate Cancer (mCRPC).

DETAILED DESCRIPTION:
This open-label, pilot trial aims to evaluate the feasibility of Sipuleucel-T given in three doses at weeks 0, 2, and 12-14; and to investigate the changes in immune response in mCRPC patients who are getting an extended course of Sipuleucel-T treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Men ≥ 18 years of age
2. Prostate cancer with history of metastasis
3. Candidates for Sipuleucel-T treatment are defined as those with asymptomatic or minimally symptomatic metastatic castrate resistant prostate cancer
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
5. Life expectancy of ≥ 6 months

Exclusion Criteria:

1. Previously received Sipuleucel-T (Provenge®)
2. Known malignancies other than prostate cancer likely to require treatment within 6 months following registration
3. A requirement for systemic immunosuppressive therapy (>10mg Prednisone daily or equivalent)
4. A history of allergic reactions attributed to compounds of similar chemical or biologic composition to Sipuleucel-T or GM-CSF
5. Any infection requiring antibiotic therapy within 1 week prior to registration

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is focused on a prostate cancer-specific group.
Enrollment: 13 (Estimated)
Dates: Start 2023-11-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients completing 3 doses of Sipuleucel-T immunotherapy. | up to 5 months
  Patients will be treated with Sipuleucel-T immunotherapy and the treatment regimen will be considered feasible if 85% of enrolled patients complete all three infusions of Sipuleucel-T treatment given at week 0, 2 and 12-14.
Proportion of subjects who have detectable elevated IgG level and/or T-cell proliferation from baseline to the follow-up of extended course of Sipuleucel-T immunotherapy. | up to 12 Months
  For patients undergoing Sipuleucel-T treatment on weeks 0, 2 and 12-14, the changes in immune response will be measured based on the detectable elevated levels of IgG and/or T-cell proliferation against various types of prostate cancer associated antigens at baseline, and at Sipuleucel-T infusion doses given at week 0, 2 and 12-14 weeks.

SECONDARY OUTCOMES:
Evaluate the mean difference in immune response to Sipuleucel-T treatment among different racial groups. | up to 12 months
  Potential difference of immune response to Sipuleucel-T immunotherapy given at weeks 0, 2 and 12-14 will be compared in patients with mCRPC of different racial groups using the one-way ANOVA or the Kruskal-Wallis test.
Evaluate the potential tumor response based on the changes in serum PSA at baseline and within 30 days of last dose. | up to 12 Months
  For patients undergoing Sipuleucel-T treatment on weeks 0, 2 and 12-14, the preliminary tumor response will be measure through the comparison of serum PSA level between baseline and within 30 days of last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Stratton, MD, Principal Investigator — Investigator
Locations (1):
- University of Oklahoma Health Sciences Center, Stephenson Cancer Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No